CLINICAL TRIAL: NCT07193290
Title: A Pilot Study to Evaluate the Expanded Reach of Decentralized Digital Skin Health Clinical Studies
Status: Completed | Type: Observational
Sponsor: Kenvue Brands LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CS2024SK100177
Record Dates: First submitted 2025-07-21; First posted 2025-09-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Skin Aging; Hair Care; Skin Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Skin Microbiome Subset: 18- to 65-year-old female subjects.
  Interventions: Other: Lifestyle Questionnaire; Other: Self-portrait image (Face and Hair)
- Skin Microbiome Subset: 18- to 65-year-old female subjects randomly assigned in the skin microbiome subset
  Interventions: Other: Lifestyle Questionnaire; Other: Self-portrait image (Face and Hair); Diagnostic Test: Skin microbiome collection

INTERVENTIONS:
Other: Lifestyle Questionnaire — All subjects will complete the lifestyle questionnaire
Other: Self-portrait image (Face and Hair) — All subjects will take one self-portrait image of their face and hair
Diagnostic Test: Skin microbiome collection — Subjects randomly assigned in the skin microbiome subset will complete the skin microbiome collection
  Groups: Skin Microbiome Subset

SUMMARY:
This is a randomized, decentralized, non-interventional clinical study. The primary objective of this study is to develop execution and efficiency metrics from completion of this study to inform on the potential design for future projects. The secondary objective of this study is to assess the main study endpoints across balanced attributes of study sub-populations.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Monk skin type 1 to 10, targeting to complete at least 100 subjects for each Monk skin type.
* 18 to 65 years old, targeting to complete:

  * 18- to 40-year-old age range: at least 50 subjects within each Monk type
  * 41- to 65-year-old age range: at least 50 subjects within each Monk type
* Lives within an Inner City, Urban, Suburban, or Rural community type (as determined by self-report or provided zip code), targeting to complete:

  * Inner City/Urban community type: at least 25 subjects within each age range and Monk type
  * Suburban/Rural community type: at least 25 subjects within each age range and Monk type
* Has electronically accepted the Consent for Photograph Release and ICD including Health Insurance Portability and Accountability Act (HIPAA) disclosure.
* Has a personal smartphone with a camera and an internet connection (wi-fi, cellular services, etc.).
* Intends to complete the study and willing and able to follow all study instructions.

Exclusion Criteria:

* Has known allergies or adverse reactions to topical adhesives.
* Is simultaneously participating in any other clinical study for the duration of this study or has participated in any product-use study within 30 days prior to remote Visit 1.
* Is an employee/contractor or immediate family member of the PI, study technology provider, laboratory, or Sponsor.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is 18- to 65-year-old, healthy female subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Interaction efficiency (contacted vs. enrolled) | 4 weeks post Last Subject's remote visit
  The number and percentage of subjects who interacted with the digital study activities vs number and percentage of subjects who completed the study.
Percent completion of subject self-taken images | 4 weeks post Last Subject's remote visit
  The number and percentage of subjects who successfully completed the self-taken images.
Percent completion of subjects participating in bio-sampling subset | 4 weeks post Last Subject's remote visit
  The number and percentage of subjects who successfully completed the bio-sampling procedures.

SECONDARY OUTCOMES:
Questionnaire results compared across skin tone | 4 weeks post Last Subject's remote visit
  The lifestyle questionnaire results will be summarized by either descriptive analysis or frequency by Monk Skin tone 1 to 10.
Questionnaire results compared across age groups | 4 weeks post Last Subject's remote visit
  The lifestyle questionnaire results will be summarized by either descriptive analysis or frequency by age groups 18- to 40-year-old and 41- to 65-year-old.

CONTACTS AND LOCATIONS:
Locations (1):
- Laina Enterprises, Inc., Apopka, Florida, United States

IPD SHARING:
Plan to Share IPD: No